CLINICAL TRIAL: NCT01163331
Title: Singing in Groups for Parkinson's Disease; A Pilot Study of Group Singing
Brief Title: Singing in Groups for Parkinson's Disease; A Pilot Study of Group Singing Therapy for PD-related Voice/Speech Impairment
Acronym: SING-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Daniel Tarsy, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000338
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Voice Quality and Voice Loudness Associated With Parkinson's Disease
Keywords: Parkinson's Disease, voice quality, vocal strength, voice loudness
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Singing Therapy Group (Experimental): Singing Therapy Group
  Interventions: Other: Singing Therapy

INTERVENTIONS:
Other: Singing Therapy — Singing therapy as a way to improve voice quality

SUMMARY:
This study will compare group singing to group speech therapy without singing. You may be eligible for this study if you have been diagnosed with PD for one year or more and you have a quiet voice or difficulty being understood.

DETAILED DESCRIPTION:
The National Parkinson Foundation Center of Excellence at Beth Israel Deaconess Medical Center is conducting a research study to test whether group singing therapy helps people with voice or speech disorders due to Parkinson's disease (PD). Communication problems, including loss of vocal loudness, affect many people with PD. While existing forms of speech therapy have been shown to be helpful, group singing may be a beneficial alternative to traditional speech therapy.

The study will involve participating in weekly treatment sessions where subjects will receive training in vocal exercises from a speech-language pathologist with expertise in PD, as well as instructions for structured home practice. Participants will be assigned to a singing or non-singing group for the 12-week treatment phase of the study. Researchers will measure subjects' vocal function and communication-related quality of life before and several times after the 12-week program. All subjects and their care partners are welcome to participate in a singing group following the study.

You may be eligible for this study if you have been diagnosed with PD for one year or more, and you have difficulty with your voice or speech such as quiet voice, or difficulty being understood.

ELIGIBILITY:
Inclusion Criteria:

* Difficulty being heard or understood
* Diagnosis of Parkinson's Disease for one year

Exclusion Criteria:

* No other neurological conditions(i.e. stroke, cerebellar ataxia) that affect voice quality
* No history of vocal chord hemorrhage

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Vocal Loudness, Vocal Quality | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.pdtrials.org